CLINICAL TRIAL: NCT05870761
Title: Phase II Trial of Combination Niraparib and Dostarlimab Therapy for Recurrent or Persistent Uterine Serous Carcinoma
Brief Title: Combination Niraparib and Dostarlimab Therapy for Recurrent or Persistent Uterine Serous Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Casey Cosgrove (Other)
Responsible Party: Sponsor-Investigator, Casey Cosgrove, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-22103; NCI-2023-03667 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Endometrial Serous Adenocarcinoma
MeSH Terms: interventions — Specimen Handling; dostarlimab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dostarlimab, niraparib) (Experimental): Patients receive dostarlimab IV and niraparib PO on study. Patients also undergo MRI/CT and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Dostarlimab; Procedure: Magnetic Resonance Imaging; Drug: Niraparib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo MRI/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Dostarlimab — Given IV
  Other Names: ANB011; Dostarlimab-gxly; Immunoglobulin G4, Anti-programmed Cell Death Protein 1 (PDCD1) (Humanized Clone ABT1 Gamma4-chain), Disulfide with Humanized Clone ABT1 Kappa-chain, Dimer; Jemperli; TSR 042; TSR-042; TSR042
Procedure: Magnetic Resonance Imaging — Undergo MRI/CT
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827

SUMMARY:
This phase II trial tests how well niraparib and dostarlimab work in treating patients with uterine serous carcinoma that has come back (after a period of improvement) (recurrent) and remains despite treatment (persistent). Niraparib belongs to a class of drugs called PARP inhibitors that prevent cancer cells from growing. Dostarlimab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Dostarlimab belongs to a class of drugs called PD-1 inhibitors that uses the patient's own immune system to treat cancer (immuno-therapy). Giving niraparib and dostarlimab may work better in treating patients with uterine serous carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy, as measured by confirmed overall response rate (ORR) (partial and complete response, PR/CR) per Response Evaluation Criteria in Solid Tumors (RECIST version [v]1.1) based on investigator assessment of the combination niraparib and dostarlimab in patients with recurrent or persistent uterine serous carcinoma (USC).

SECONDARY OBJECTIVES:

I. Estimate the progression-free survival (PFS). II. Estimate clinical benefit rate (CBR), defined as the percentage of patients who have achieved complete response (CR), partial response (PR) or stable disease (SD).

III. Evaluate the safety and tolerability of niraparib and dostarlimab combination.

TRANSLATIONAL OBJECTIVE:

I. Biomarker evaluation to predict response.

OUTLINE:

Patients receive dostarlimab intravenously (IV) and niraparib orally (PO) on study. Patients also undergo magnetic resonance imaging (MRI)/computed tomography (CT) and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 6 months for 2 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have recurrent or persistent uterine serous carcinoma based on previous biopsy or surgery, and have previously received at least carboplatin/paclitaxel. Mixed and carcinosarcoma histology cases will be eligible if there is a serous component in the tumor
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Participant must be >= 18 years of age
* Patient has archival tumor tissue available or a fresh biopsy of recurrent or persistent tumor must be obtained prior to study treatment initiation
* Patient must have measurable disease by RECIST
* No more than three prior chemotherapy regimens (does not include chemoradiation) are permitted. One of the previous lines of treatment must include carboplatin and paclitaxel
* Prior PD1/PDL1 inhibitors (including single-agent pembrolizumab, other immunotherapy agents, or combination pembrolizumab and lenvatinib) therapy will be allowed if the patient did not have immune associated toxicity leading to discontinuation.

  * Patients who have progressed on prior PD1/PDL1 inhibitors may be allowed to participate if the study PI and treating physician deem it to be within the patient's best interest.
* Prior chemoradiation therapy for adjuvant treatment or pelvic recurrence is permitted. Chemotherapy in this setting, is not counted as prior line of chemotherapy
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance >= 60 mL/min using the Cockcroft-Gault equation
* Total bilirubin =< 1.5 x ULN (=< 2.0 in patients with known Gilberts syndrome) OR direct bilirubin =< 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase =< 2.5 x ULN unless liver metastases are present, in which case they must be =< 5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy and dose < 10 mg of prednisone or equivalent
* Participant must be able to take oral medications
* Participant must agree to not donate blood during the study or for 120 days after the last dose of study treatment
* If of childbearing potential, has a negative serum pregnancy test within 7 days prior to taking study medication and agrees to abstain from activities that could result in pregnancy from enrollment through 180 days (6 months) after the last dose of study treatment or be of non-childbearing potential. Non childbearing potential is defined as follows (by other than medical reasons):

  * >= 45 years of age and has not had menses for > 1 year
  * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Surgically sterile as defined as post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient
* Participant must agree to not breastfeed during the study or for 120 days after the last dose of study treatment
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent
* Must have recovered to =< grade 1 from all toxicities related to prior treatment that are deemed clinically relevant in the opinion of the investigator at time of enrollment

Exclusion Criteria:

* Participant must not be simultaneously enrolled in any interventional clinical trial
* Participant must not have had major surgery =< 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects
* Participant must not have received investigational therapy =< 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior initiating protocol therapy
* Participant's last treatment with platinum based chemotherapy was =< 4 weeks from initiation of protocol therapy
* Participant has had radiation therapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to day 1 of protocol therapy
* Participant must not have a known hypersensitivity to niraparib and dostarlimab components or excipients
* Participant must not have previously progressed on PARP inhibitor
* Participant experienced >= grade 3 immune-related adverse event (AE) with prior immunotherapy, with the exception of non-clinically significant lab abnormalities
* Participant must not have received a transfusion (platelets or red blood cells) =< 4 weeks prior to initiating protocol therapy
* Participant must not have received colony-stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy
* Participant has had any known grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment
* Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled hypertension, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent. Participants with hypertension but be well controlled before first dose of niraparib
* Participant must not have had diagnosis, detection, or treatment of another type of cancer =< 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
* Participant must not have a known history of brain or leptomeningeal metastases
* Participant has a diagnosis of immunodeficiency or has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy
* Participant has a known history of human immunodeficiency virus (type 1 or 2 antibodies)
* Participant has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected)
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement hormone therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not an exclusion criterion
* Participant must not have a history of interstitial lung disease
* Participant is considered a poor medical risk that would interfere with cooperation with the requirements of the study
* Participant has received a live vaccine within 30 days of initiating protocol therapy
* Participant has a history of posterior reversible encephalopathy syndrome (PRES)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years
  Defined as the percentage of patients with complete response (CR), or partial response (PR), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v.) 1.1 criteria using investigator's review. Will be estimated and reported with 95% confidence intervals (exact).

SECONDARY OUTCOMES:
Clinical benefit rate | Up to 2 years
  Clinical benefit rate (CR, PR, or stable disease [SD]) by RECIST v1.1 will be also estimated and reported with 95% confidence interval (exact).
Progression free survival (PFS) | From the date of study entry until disease progression or death (whichever occurs first), assessed up to 2 years
  PFS will be analyzed by Kaplan-Meier (KM) methods, and point estimates and 2-sided 95% confidence intervals for PFS will be reported for selected times such as 3, 6 and 12 months from treatment start using Greenwood's variance and the log-log transform method. Median PFS time, if attained, will also be reported.
Overall survival (OS) | Up to 2 years
  OS will be analyzed by KM methods. Median OS time, if attained, will also be reported.
Duration of response (DoR) | Up to 2 years
  DoR will be evaluated by restricted mean DoR.
Incidence of adverse events (AEs) | Up to 90 days
  Toxicity will be summarized by reporting the number of patients treated, the number who experience treatment related toxicity, serious adverse events and grade 3 or higher AE, the number of patients who discontinue therapy, and the reasons for discontinuation. Comprehensive safety data on all grade 3 and 4 toxicities will be tabulated by type, grade, and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Cosgrove, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu